CLINICAL TRIAL: NCT02114385
Title: A Randomized, Double-Blinded, Controlled With GARDASIL (Human Papillomavirus Vaccine [HPV] [Types 6, 11, 16, 18] (Recombinant, Adsorbed)), Phase 3 Clinical Trial to Study the Immunogenicity and Tolerability of V503 (9-Valent Human Papillomavirus L1 Virus-Like Particle [VLP] Vaccine) in 16- to 26-year-old Men
Brief Title: A Study to Compare Immune Response of V503 to Gardasil in 16- to 26-year-old Men (V503-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V503-020; 2013-003399-10 (EudraCT Number); GDS07C (Other: MCMVaccBV (SPMSD) Protocol Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Papilloma Viral Infection
Keywords: Prevention
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- V503 (Experimental): 9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine, 0.5-mL intramuscular injection in 3 dose regimen at Day 1, Month 2, and Month 6
  Interventions: Biological: V503
- GARDASIL (Active Comparator): Quadrivalent HPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine, 0.5-mL intramuscular injection in 3 dose regimen at Day 1, Month 2, and Month 6
  Interventions: Biological: GARDASIL

INTERVENTIONS:
Biological: V503 — 9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine, 0.5-mL intramuscular injection
  Other Names: 9vHPV vaccine
  Arms: V503
Biological: GARDASIL — Quadrivalent HPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine, 0.5-mL intramuscular injection
  Other Names: qHPV vaccine
  Arms: GARDASIL

SUMMARY:
Primary objective

To demonstrate that administration of V503 induces non-inferior Geometric Mean Titres (GMTs) for serum anti-HPV 6, 11, 16, and 18, compared to GARDASIL in 16- to 26-year-old men

DETAILED DESCRIPTION:
Secondary objectives

* To evaluate the tolerability of V503 in 16- to 26-year-old men.
* To summarise humoral immune responses, including anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, 58 GMTs and seroconversion rates at 4 weeks post-dose 3, in 16- to 26-year-old men who received V503 or GARDASIL

ELIGIBILITY:
Inclusion Criteria:

* Subject is a man, between the ages of 16 years and 0 days and 26 years and 364 days on the day of enrolment.
* Subject is a man who has had no more than 5 lifetime female sexual partners.
* Subject is judged to be in good physical health on the basis of medical history, physical examination, and laboratory results.
* Subject, or subject's parent or guardian, fully understand study procedures, alternative treatments available, the risks involved with the study, and voluntarily agree to participate by giving written informed consent.

Exclusion Criteria:

* Subject who has had sex with a male partner.
* Subject has a history of HPV-related external genital lesions or HPV-related anal lesions
* Subject has a known allergy to any vaccine component, including aluminium, yeast, or BENZONASE
* Subject has a history of severe allergic reaction that required medical intervention.
* Subject has thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Subject is concurrently enrolled in clinical studies of investigational medicinal products.
* Subject has donated blood within 1 week prior to the Day 1 vaccination, or intends to donate during Day 1 through Month 7 of the study.
* Subject is currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Subject has had a splenectomy.
* Subject is receiving or has received in the year prior to enrolment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide, TNF-α antagonists, monoclonal antibody therapies, intravenous gamma globulin, antilymphocyte sera, or other therapy known to interfere with the immune response.
* Subject has received any immune globulin product or blood-derived product within the 6 months prior to the Day 1 vaccination, or plans to receive any such product during Day 1 through Month 7 of the study.
* Subject has received non-replicating (inactivated) vaccines within 14 days prior to the Day 1 vaccination or has received replicating (live) vaccines within 21 days prior to the Day 1 vaccination.
* Subject has received a marketed HPV vaccine, or has participated in an HPV vaccine clinical trial and has received either active agent or placebo.
* Subject has had a fever within the 24-hour period prior to the Day 1 vaccination.
* Subject has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.
* Subject is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
* Subject is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug abuse or dependence. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems as a result of alcohol use.
* Subject, or subject's parent or guardian, is or has an immediate family member (spouse or children) who is investigational site or sponsor staff directly involved with this trial.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2014-03-24; Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- Belgium (3):
  - Sanofi Pasteur MSD Investigational Site 1002, Ghent
  - Sanofi Pasteur MSD Investigational Site 1003, Leuven
  - Sanofi Pasteur MSD Investigational Site 1001, Wilrijk
- Sanofi Pasteur MSD Investigational Site 3001, Mainz, Germany
- Netherlands (3):
  - Sanofi Pasteur MSD Investigational Site 4001, Amsterdam
  - Sanofi Pasteur MSD Investigational Site 4003, Amsterdam
  - Sanofi Pasteur MSD Investigational Site 4002, Nijmegen

REFERENCES:
- [Result] Van Damme P, Meijer CJLM, Kieninger D, Schuyleman A, Thomas S, Luxembourg A, Baudin M. A phase III clinical study to compare the immunogenicity and safety of the 9-valent and quadrivalent HPV vaccines in men. Vaccine. 2016 Jul 29;34(35):4205-4212. doi: 10.1016/j.vaccine.2016.06.056. Epub 2016 Jun 25. PMID 27354258
- [Derived] Moreira ED, Giuliano AR, de Hoon J, Iversen OE, Joura EA, Restrepo J, Van Damme P, Vandermeulen C, Ellison MC, Krick A, Shields C, Heiles B, Luxembourg A. Safety profile of the 9-valent human papillomavirus vaccine: assessment in prior quadrivalent HPV vaccine recipients and in men 16 to 26 years of age. Hum Vaccin Immunother. 2018 Feb 1;14(2):396-403. doi: 10.1080/21645515.2017.1403700. Epub 2017 Dec 14. PMID 29211620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 502 participants were screened and 500 were randomized
Period: Overall Study
Arm/Group | V503 | GARDASIL
Started | 249 | 251
Vaccinated | 249 | 251
Completed | 246 | 243
Not Completed | 3 | 8
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 6

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | V503 | GARDASIL | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.8 (2.7) | 21.3 (3.0) | 21.0 (2.8)
Age, Customized [Number; unit: Participants]
  <18 years old | 37 | 38 | 75
  >=18 years old | 212 | 213 | 425
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 249 | 251 | 500

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) to HPV Types 6/11/16/18
Description: Serum antibodies to HPV types 6, 11, 16, and 18 were measured with a Competitive Luminex Immunoassay. Titers are reported in milli Merck Units/mL.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: All randomized participants. The number contributing to each data point is participants who received all 3 vaccinations within acceptable day ranges, had Month 7 serology for the HPV type within acceptable day ranges, were seronegative at Day 1, and had no protocol violations that interfered with evaluation of immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 249 | 251
milli Merck U/mL
  HPV Type 6: number analyzed (Participants) | 228 | 226
  HPV Type 6 | 758.3 [665.9 to 863.4] | 618.4 [554.0 to 690.3]
  HPV Type 11: number analyzed (Participants) | 228 | 226
  HPV Type 11 | 681.7 [608.9 to 763.4] | 769.1 [683.5 to 865.3]
  HPV Type 16: number analyzed (Participants) | 234 | 237
  HPV Type 16 | 3924.1 [3513.8 to 4382.3] | 3787.9 [3378.4 to 4247.0]
  HPV Type 18: number analyzed (Participants) | 234 | 236
  HPV Type 18 | 884.3 [766.4 to 1020.4] | 790.9 [683.0 to 915.7]
Statistical Analysis 1: Comparison: V503 vs GARDASIL; HPV Type 6; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.50; p < 0.001, ANOVA; GMT Ratio = 1.23, 95% CI 2-sided [1.04 to 1.45] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 2: Comparison: V503 vs GARDASIL; HPV Type 11; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.50; p < 0.001, ANOVA; GMT Ratio = 0.89, 95% CI 2-sided [0.76 to 1.04] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 3: Comparison: V503 vs GARDASIL; HPV Type 16; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.50; p < 0.001, ANOVA; GMT Ratio = 1.04, 95% CI 2-sided [0.89 to 1.21] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 4: Comparison: V503 vs GARDASIL; HPV Type 18; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.50; p < 0.001, ANOVA; GMT Ratio = 1.12, 95% CI 2-sided [0.91 to 1.37] — GMT ratio = GMT (V503) / GMT (Gardasil)

2. Secondary Outcome: GMTs to HPV Types 31/33/45/52/58
Description: Serum antibodies to HPV types 31, 33, 45, 52, and 58 were measured with a Competitive Luminex Immunoassay. Titers are reported in milli Merck Units/mL.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck U/mL
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 249 | 251
milli Merck U/mL
  HPV Type 31: number analyzed (Participants) | 234 | 237
  HPV Type 31 | 794.4 [694.2 to 909.2] | 14.8 [12.5 to 17.5]
  HPV Type 33: number analyzed (Participants) | 236 | 236
  HPV Type 33 | 460.5 [410.6 to 516.4] | 3.4 [3.1 to 3.7]
  HPV Type 45: number analyzed (Participants) | 232 | 236
  HPV Type 45 | 262.9 [226.2 to 305.5] | 2.5 [2.3 to 2.8]
  HPV Type 52: number analyzed (Participants) | 235 | 236
  HPV Type 52 | 430.7 [377.8 to 491.0] | 1.9 [1.8 to 2.1]
  HPV Type 58: number analyzed (Participants) | 232 | 233
  HPV Type 58 | 691.0 [614.9 to 776.5] | 5.7 [5.0 to 6.5]

3. Secondary Outcome: Percentage of Participants Who Are Seropositive for HPV Types 6/11/16/18/31/33/45/52/58
Description: Serum antibodies to HPV types were measured with a Competitive Luminex Immunoassay. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30; HPV Type 11: ≥16; HPV Type 16: ≥20; HPV Type 18: ≥24; HPV Type 31: ≥10; HPV Type 33: ≥8; HPV Type 45: ≥8; HPV Type 52: ≥8; HPV Type 58: ≥8.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 249 | 251
Percentage of participants
  HPV Type 6: number analyzed (Participants) | 228 | 226
  HPV Type 6 | 98.2 [95.6 to 99.5] | 98.7 [96.2 to 99.7]
  HPV Type 11: number analyzed (Participants) | 228 | 226
  HPV Type 11 | 100 [98.4 to 100] | 100 [98.4 to 100]
  HPV Type 16: number analyzed (Participants) | 234 | 237
  HPV Type 16 | 100 [98.4 to 100] | 100 [98.5 to 100]
  HPV Type 18: number analyzed (Participants) | 234 | 236
  HPV Type 18 | 99.6 [97.6 to 100] | 99.6 [97.7 to 100]
  HPV Type 31: number analyzed (Participants) | 234 | 237
  HPV Type 31 | 100 [98.4 to 100] | 61.6 [55.1 to 67.8]
  HPV Type 33: number analyzed (Participants) | 236 | 236
  HPV Type 33 | 100 [98.4 to 100] | 16.9 [12.4 to 22.4]
  HPV Type 45: number analyzed (Participants) | 232 | 236
  HPV Type 45 | 100 [98.4 to 100] | 9.3 [5.9 to 13.8]
  HPV Type 52: number analyzed (Participants) | 235 | 236
  HPV Type 52 | 100 [98.4 to 100] | 2.5 [0.9 to 5.5]
  HPV Type 58: number analyzed (Participants) | 232 | 233
  HPV Type 58 | 100 [98.4 to 100] | 36.1 [29.9 to 42.6]

4. Secondary Outcome: Percentage of Participants With One or More Adverse Events
Description: The percentage of participants with one or more adverse events was assessed.
Time Frame: Up to 15 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 82.3 [76.9 to 86.8] | 81.9 [76.5 to 86.4]

5. Secondary Outcome: Percentage of Participants With Study Discontinuation Due to an Adverse Event
Description: The percentage of participants discontinued from the study due to an adverse event was assessed.
Time Frame: Up to Month 7
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 0 [0 to 1.5] | 0 [0 to 1.5]

6. Secondary Outcome: Percentage of Participants With One or More Injection-site Adverse Reactions
Description: The percentage of participants with one or more injection-site adverse reactions (solicited or unsolicited) was assessed.
Time Frame: Up to 5 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 79.0 [73.4 to 83.9] | 72.2 [66.2 to 77.7]

7. Secondary Outcome: Percentage of Participants With Maximum Temperature ≥37.8 °C
Description: The percentage of participants with a maximum temperature ≥37.8 °C was assessed.
Time Frame: Up to 5 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 2.8 | 2.4

8. Secondary Outcome: Percentage of Participants With One or More Systemic Adverse Events
Description: The percentage of participants with one or more systemic adverse events was assessed.
Time Frame: Up to 15 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 40.7 [34.6 to 47.1] | 40.3 [34.2 to 46.7]

9. Secondary Outcome: Percentage of Participants With One or More Serious Adverse Events
Description: The percentage of participants with one or more serious adverse events was assessed.
Time Frame: Up to 15 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 248 | 248
Percentage of participants | 0.0 [0.0 to 1.5] | 0.0 [0.0 to 1.5]

ADVERSE EVENTS:
Time Frame: All adverse events: up to 15 days after each vaccination; serious adverse events: up to Month 7
Arm/Group | V503 | GARDASIL
Serious Adverse Events (participants affected / at risk) | 0/248 | 6/248
Other Adverse Events (participants affected / at risk) | 196/248 | 189/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=248) | GARDASIL (N=248)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=248) | GARDASIL (N=248)
Injection-site erythema (General disorders) | 38 (62) | 43 (64)
Injection-site pain (General disorders) | 193 (443) | 174 (350)
Injection-site swelling (General disorders) | 36 (47) | 23 (35)
Nasopharyngitis (Infections and infestations) | 11 (13) | 14 (16)
Headache (Nervous system disorders) | 29 (43) | 37 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.